CLINICAL TRIAL: NCT03176147
Title: Clinical and Biological Predictive Factors of Iron Deficiency Anemia in the Third Trimester of Pregnancy
Brief Title: Iron Metabolism Parameters At First Trimester and preGnancy outcomE
Acronym: IMAGE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-336; 2015-A00454-45 (Other: 2015-A00454-45)
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Iron Deficiency Anemia
Keywords: Anemia; Pregnancy; Hepcidine; Iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women are included during the ultrasound of T1. Written consent will be sought after delivery of the information notice.
  Interventions: Other: Iron deficiency anemia

INTERVENTIONS:
Other: Iron deficiency anemia — The prevalence of iron deficiency anemia is determined at T3 (after 34 SA). The predictive factors for this anemia will be sought according to the data collected in T1.

SUMMARY:
Iron deficiency anemia is the leading cause of anemia during pregnancy, which can still reach 10 to 20% of pregnant women in developed countries, with potentially serious consequences for the child. Systematic iron supplementation remains controversial.

This study aims to identify in the first trimester of pregnancy clinical and biological predictive factors for the occurrence of iron deficiency anemia in the third trimester of pregnancy.

DETAILED DESCRIPTION:
Objectives: The main objective is to determine the prevalence of anemia (Hb ≤ 11 g / dl) in the third trimester of pregnancy (T3) and to identify the predictive factors in the first trimester (T1).

Type of study: Prospective monocentric cohort.

Experimental plan: Pregnant women are included during the ultrasound of T1. Written consent will be sought after delivery of the information notice. Hemoglobin, classical iron balance (ferritin, transferrin saturation coefficient) as well as other original parameters: hepcidin and the soluble transferrin receptor are assayed. Socioeconomic and clinical parameters likely to favor an iron deficiency are sought through validated questionnaires. Nutritional advice, combined with martial supplementation if necessary, is given according to a standardized management protocol resulting from the current international recommendations and validated by an internal committee. The prevalence of iron deficiency anemia is determined at T3 (after 34 SA). The predictive factors for this anemia will be sought according to the data collected in T1.

The 2012 WHO's recommendations are in favour of a systematic supplementation of pregnant women. Epidemiological studies show that the anaemia at the end of pregnancy increases the risk of severe anaemia in the postpartum hospital stay and the frequency of transfusions in the mother is multiplied by 9. The quality of life of the mother seems too altered by the anaemia with increased susceptibility to infections, cognitive and emotional disorders in the postpartum period and a decrease of capacity of work and performance. In the human new-born, the anaemia is associated with a risk of prematurity, low weight birth and especially a certain degree of later psycho-motor delay, or even perinatal mortality. Side effects of iron orally, it's cost, make debatable systematic supplementation as interventional studies have given contradictory results in terms of morbidity and mortality infant. In areas where the anaemia prevalence is very high, a systematic supplementation of pregnant by 60 mg of iron (with folic acid) is beneficial in children on clues of psycho-intellectual development at 12, 18 and 24 months while multiple supplementation in micronutrients (containing 30 mg of iron) is not effective. However, systematic supplementation in countries with high socioeconomic level did debate. An Australian study Interventional, controlled, randomized conducted at 430 women showed no efficacy on the intellectual development of children in 4 years, without changing the quality of life of the mother during pregnancy, the authors observing even an increase of abnormal behaviors of the children of the mothers in the Group supplemented iron. In another study, the rational is highly questionable, a treatment by Iron versus placebo was given to pregnant women not anaemic with a high haemoglobin (an average of 14 g/dl): the women who took iron had high blood pressure at the end of pregnancy more and their children had a lower birth for the term weight.

In a developed country such as the France, one can legitimately wonder about the potentially harmful effects of routine iron supplementation for a population of pregnant women mainly not anaemic. In Great Britain of the recently published recommendations are pronounced against a systematic supplementation of iron in pregnant women. Other European authors advocate focused on the rate of ferritin supplementation. However, we are lacking of studies allowing, from clinical criteria and biological precise, to better target pregnant women who could benefit from supplementation of iron in the first quarter.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the first trimester between 11SA and 13 SA + 6 days
* A written agreement is needed

Exclusion Criteria:

* Women who do not know enough about reading and writing French to answer questionnaires
* Women under 15 at inclusion

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The women were screened at the maternity clinic of the gynecology-obstetrics department of CHU Estaing in Clermont-Ferrand, France.
Sampling Method: Non-Probability Sample
Enrollment: 865 (Estimated)
Dates: Start 2015-11-12 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin value | in the third trimestry of pregnancy

SECONDARY OUTCOMES:
Rate of clinical and biological factors per patient | at the first trimestry of pregnancy
  demographics and clinical factors and biological factors (hepcidine, ferritine, RST)
Rate of demographics and clinical factors per patient | at the first trimestry of pregnancy
  biological factors (hepcidine, ferritine, RST)
Rate of biological factors per patient | at the first trimestry of pregnancy
  Such as : hepcidine, ferritine, RST

CONTACTS AND LOCATIONS:
Overall Officials: Marc RUIVARD, MD, PhD, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France